CLINICAL TRIAL: NCT06576011
Title: 2 College Truths and 1 Lie: Social Media Embedded Gamified Normative Re-education
Brief Title: 2 College Truths and 1 Lie
Acronym: 2T1L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola Marymount University (Other)
Responsible Party: Principal Investigator, Dr. Joseph LaBrie, Professor of Psychology, Loyola Marymount University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R34AA030139-02 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Underage Drinking
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study conditions are randomly assigned and the intervention delivery is automated through digital advertisements on social media. Senior members of the research team will have a record of the participants randomized to each condition, but the delivery of intervention content is automated. Junior members of the research team responsible for sending follow-up survey reminders will not be aware of participant condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gamified Social Norms Marketing Campaign (Experimental): Participants randomized to this arm will receive a gamified social norms marketing campaign that is primarily delivered via advertisements on the social media platform Instagram.
  Interventions: Behavioral: Gamified Social Norms Marketing Campaign
- Social Norms Marketing Campaign (Experimental): Participants randomized to this arm will receive a social norms marketing campaign that is primarily delivered via advertisements on the social media platform Instagram.
  Interventions: Behavioral: Social Norms Marketing Campaign
- Assessment-Only Control (No Intervention): Participants do not receive anything besides the surveys.

INTERVENTIONS:
Behavioral: Gamified Social Norms Marketing Campaign — This intervention is a gamified social norms marketing campaign (SNMC) primarily disseminated via advertisements on Instagram. These advertisements will invite students to participate in a game about student life at their university, during which misperceived alcohol norms will be corrected. The gamified SNMC spans the first full six weeks of students' first fall semester in college and includes three rounds of play. Round one occurs during the first two weeks, round two during the third and fourth weeks, and round three during the fifth and sixth weeks. In the game, participants are asked to identify whether normative facts related to a variety of topics are true or false. Correct feedback is then provided, intended to reinforce accurate norms related to alcohol use, which are embedded alongside other facts about college life.
  Arms: Gamified Social Norms Marketing Campaign
Behavioral: Social Norms Marketing Campaign — This intervention is a social norms marketing campaign that is primarily delivered via advertisements on Instagram. These advertisements will contain normative facts related to student life at their university, during which misperceived alcohol norms will be corrected.
  Arms: Social Norms Marketing Campaign

SUMMARY:
This pilot randomized control trial (RCT) aims to assess the feasibility and efficacy of 2 College Truths & 1 Lie (2T1L), a gamified social norms marketing campaign (SNMC) aimed at preventing and reducing first-year college student drinking. This program is designed to correct overestimations of peers' alcohol use behaviors, which, as shown in previous research, influence one's own future drinking behaviors. To examine the efficacy of 2T1L, this pilot trial will use a longitudinal design to determine whether playing 2T1L during the first few weeks of college will prevent increases in drinking or reduce subsequent alcohol use among first-year students during the same year, relative to exposure to a static social media-delivered SNMC or an assessment-only control condition. The investigators hypothesize that students randomized to receive the interactive 2T1L SNMC game will report less state psychological reactance in response to normative campus drinking statistics than students randomized to the non-gamified SNMC condition. Further, students in the 2T1L game condition will report greater accuracy in their perceptions of campus drinking norms and consume less alcohol following the six-week SNMC (short-term follow-up) and toward the end of the first year (long-term follow-up) compared to those randomized to both the active non-gamified SNMC and assessment-only control conditions.

DETAILED DESCRIPTION:
A pilot RCT will be conducted to evaluate the feasibility and efficacy of the proposed gamified normative re-education campaign, 2 College Truths & 1 Lie (2T1L), which will be embedded on the most popular social media platforms associated with high-risk drinking during the first year of college. Incoming first-year students will be invited to participate in an online survey during the month prior to the start of the fall semester to determine baseline drinking norms and alcohol use. An automated randomizer will be programmed into the online survey to non-visibly assign participants to the intervention (n=138), active control (n=138), or assessment-only control (n=138) group. On the first day of the second week of classes, ads promoting participation in the gamified and static versions of 2T1L will begin to appear in the Instagram accounts of participants randomized to the intervention and active control conditions, respectively. These ads will continue to run over the course of the first six weeks, with a new ad promoting the current round of play every two weeks. Approximately one month following the conclusion of the final round of play, participants in all three conditions will be invited to complete the first follow-up survey (short-term intervention effects), which will include the same measures of drinking norms and alcohol use assessed at baseline. Six months post-intervention, participants will be invited to complete a second follow-up survey to assess the long-term effects of the intervention. At both the 1-month and 6-month follow-ups, the investigators expect that participants randomized to the intervention group will report greater accuracy in their perceptions of campus drinking norms and consume less alcohol relative to those randomized to both the active non-gamified SNMC and assessment-only control conditions.

ELIGIBILITY:
Inclusion Criteria:

* Incoming first-year student with valid LMU email address
* 18-20 years of age
* Checks their Instagram 1-3+ times per week
* Consented to participate in the study

Exclusion Criteria:

* Not an incoming first year student attending LMU
* Under 18 years of age or over 20 years of age
* Do not have an Instagram account or checks it fewer than 1-3+ times per week
* Did not consent to participate in the study

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 392 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Daily Drinking at 4 Months | baseline, 4 months
  Self-reported number of drinks consumed during an average week in the past 30 days.
Change from Baseline Daily Drinking at 9 Months | baseline, 9 months
  Self-reported number of drinks consumed during an average week in the past 30 days.
Change from Peak Drinking Occasion at 4 Months | baseline, 4 months
  Self-reported max number of drinks consumed on a single occasion in the past 30 days.
Change from Baseline Peak Drinking Occasion at 9 Months | baseline, 9 months
  Self-reported max number of drinks consumed on a single occasion in the past 30 days.
Change from Baseline Descriptive Peer Drinking Norms- Drinking Norms Rating form at 4 Months | baseline, 4 months
  Assesses perceptions of weekly alcohol consumption among peers over the past 30 days.
Change from Baseline Descriptive Peer Drinking Norms- Drinking Norms Rating form at 9 Months | baseline, 9 months
  Assesses perceptions of weekly alcohol consumption among peers over the past 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola Marymount University, Los Angeles, California, United States